CLINICAL TRIAL: NCT04606875
Title: Assessment of Campbell Score as a Means of Predicting Suicidal Ideation High Risk Patients
Brief Title: Correlation of Campbell Score With Suicidal Ideation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Therapeutic Solutions International (Industry)
Responsible Party: Sponsor
Other Study IDs: Campbell Neuro 001
Record Dates: First submitted 2020-10-22; First posted 2020-10-28 (Actual); Last update posted 2020-10-28 (Actual); Status verified 2020-10

CONDITIONS: Suicidal Ideation
Keywords: interleukin-6, suicidal ideation, immunology
MeSH Terms: conditions — Suicidal Ideation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Control Group: Subjects will have no personal or family psychiatric history and no suicide attempts.
  Interventions: Diagnostic Test: Campbell Score
- Patients with Suicidal Ideation and Low Acquired Capability: Subjects will have suicidal ideation (Hamilton Depression Rating Scale suicide item >2) and reported low acquired capability for suicide (Acquired Capability for Suicide Scale <20)
  Interventions: Diagnostic Test: Campbell Score
- Patients with Suicidal Ideation and High Acquired Capability: Subjects will have suicidal ideation (Hamilton Depression Rating Scale suicide item >2) and reported high acquired capability for suicide (Acquired Capability for Suicide Scale >60)
  Interventions: Diagnostic Test: Campbell Score

INTERVENTIONS:
Diagnostic Test: Campbell Score — The Campbell Score is a blood based assessment of inflammatory and immunologically associated markers that is currently in development as a means of predicting suicidal ideations.

SUMMARY:
The Campbell Score is a blood based means of assessing molecules believed to be associated with suicidal ideation and in some cases successful suicide.

The current clinical trial will assess the Campbell Score in 3 groups:

Group 1: 10 patients with no personal or family psychiatric history and no suicide attempts.

Group 2: 10 patients with suicidal ideation (Hamilton Depression Rating Scale suicide item >2) and reported low acquired capability for suicide (Acquired Capability for Suicide Scale <20).

Group 3: 10 patients with suicidal ideation (Hamilton Depression Rating Scale suicide item >2) and reported high acquired capability for suicide (Acquired Capability for Suicide Scale >60).

The goal of the study is to confirm efficacy of Campbell Score in identifying patients with high suicidal ideation potential.

ELIGIBILITY:
Inclusion Criteria:

* Capability of giving informed consent
* Agree to abide by the study protocol and its restrictions and be able to complete all aspects of the study.
* Be diagnosed with Suicide ideation/attempts/gestures

Exclusion Criteria:

- Not currently pregnant or lactating (due to potential confounding of brain activity as a result of differing hormone levels)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will comprise of 10 healthy volunteers, as well as 20 patients with suicidal ideations. 10 of the patients will have low acquired capability for suicide, and 10 will have high acquired capability for suicide.
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2020-11-05 (Estimated); Primary Completion 2021-01-13 (Estimated); Study Completion 2021-02-13 (Estimated)

PRIMARY OUTCOMES:
Assessment of Campbell Score | 1 week to compare the records with the Campbell Score
  Campbell Score will be compared between healthy volunteers, patients with suicidal idea with low acquired capability for suicide, and patients with suicidal idea with high acquired capability for suicide.
Assessment of Correlation between Campbell Score and Beck Scale for Suicidal Ideation | 1 week to compare the records with the Campbell Score
  Campbell Score will be compared to scoring of patients on the Beck Scale for Suicidal Ideation

CONTACTS AND LOCATIONS:
Locations (1):
- Therapeutic Solutions International, Oceanside, California, United States

IPD SHARING:
Plan to Share IPD: Undecided